CLINICAL TRIAL: NCT05184686
Title: Effects of Electromagnetic Field and Noise on Alpha Band and Functional Connections of Human Resting Electroencephalogram
Brief Title: Effects of Electromagnetic Field and Noise on Resting Electroencephalogram of Health Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KY20212098-F-1
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2021-12

CONDITIONS: Electroencephalography; Electromagnetic; Noise Exposure
Keywords: Electroencephalography; Noise Exposure; electromagnetic Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- noise(low-level) and RF(low-level) (Active Comparator)
  Interventions: Other: noise expose; Other: RF expose
- noise(high-level) and RF(low-level) (Active Comparator)
  Interventions: Other: noise expose; Other: RF expose
- noise(high-level) and RF(high-level) (Active Comparator)
  Interventions: Other: noise expose; Other: RF expose
- noise(low-level) and RF(high-level) (Active Comparator)
  Interventions: Other: noise expose; Other: RF expose

INTERVENTIONS:
Other: noise expose — simulate noise expose environments
Other: RF expose — simulate RF expose environments

SUMMARY:
With the development of science and technology, there are more and more electromagnetic and noise factors in the working and living environment. These two factors often exist together, and their impact on people may interact. Scalp EEG is a classic nerve detection technology, which can reflect the functional state of the brain in a non-invasive and real-time manner. This project intends to use EEG technology to study the effects of electromagnetism and noise on human brain function.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-30 years old, right-handed, with normal hearing and normal visual or corrected acuity;

Exclusion Criteria:

* Have history of smoking, alcohol abuse, no history of neurological or psychiatric disorders (e.g., epilepsy), no relevant family history, and no recent medication use;
* Have history of surgery for head injury, no metal implants in the body (including braces);
* Sleep-wake time irregular， with sleep disturbance;
* Have history of noise allergy;
* Participate in similar psychological experiments during 2 months.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
alpha band power of the EEG spectral | Procedure (record EEG during the noise and RF expose, and then compute the alpha band power of the EEG )
theta band power/beta band power of the EEG spectral | Procedure (record EEG during the noise and RF expose, and then compute theta/beta of the EEG )

CONTACTS AND LOCATIONS:
Locations (1):
- Air Force Military Medical University, Xi’an, Shanxi, China